CLINICAL TRIAL: NCT07264881
Title: A Prospective, Longitudinal, Multi-modal Study Evaluating the Utility of Acute Phase UFR (IVUS-FFR) to Predict Functional Significance in the Stable Phase for Patients With Acute Coronary Syndrome (ACS)
Brief Title: For Patients With Myocardial Infarction and Multiple Vessel: Testing if Ultrasound (UFR) Can Guide All Needed Treatment in One Procedure, Avoiding a Return Hospital Visit for a Second Operation.
Acronym: ACT-EVOLVE
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Hai Gao, Chief Physician, Beijing Anzhen Hospital
Other Study IDs: KS2025241; KS2025241 (Other: BeijingAnzhen)
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Microvascular Obstruction (MVO); Multivessel Coronary Artery Disease; ACS (Acute Coronary Syndrome); ST Elevation Myocardial Infarction (STEMI)
Keywords: Acute Coronary Syndrome; Fractional Flow Reserve,; Intravascular Ultrasound; Virtual Fractional Flow Reserve; Functional Drift; Coronary Microvascular Dysfunction; Index of Microcirculatory Resistance; Non-Culprit Vessel; ST Elevation Myocardial Infarction; Non-ST Elevation Myocardial Infarction; Cardiac Magnetic Resonance; Microvascular Obstruction; Staged Revascularization; Computational Fluid Dynamics
MeSH Terms: conditions — Acute Coronary Syndrome; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- ACS with MVD Cohort: A single prospective, observational cohort of 200 patients presenting with Acute Coronary Syndrome (ACS) and multi-vessel disease (MVD). This single cohort will be pre-stratified at enrollment into two groups for comparative analysis: 1) STEMI (N≈100) and 2) High-Risk NSTEMI (N≈100). All participants undergo the identical longitudinal assessment.
  Interventions: Diagnostic Test: IVUS-based Fractional Flow Reserve (UFR); Diagnostic Test: Invasive Coronary Physiology Measurement (FFR/RFR/IMR); Diagnostic Test: Cardiac Magnetic Resonance (CMR)

INTERVENTIONS:
Diagnostic Test: IVUS-based Fractional Flow Reserve (UFR) — UFR is a "virtual" fractional flow reserve calculated from Intravascular Ultrasound (IVUS) images using computational fluid dynamics.
  In this study, it is calculated from IVUS runs of the Non-Culprit Vessel (NCV) performed at the T0 (Acute) procedure. This T0 UFR value is the primary diagnostic test being evaluated against the T1 (30-day) pFFR gold standard. UFR will also be assessed at the T2 (1-year) follow-up.
Diagnostic Test: Invasive Coronary Physiology Measurement (FFR/RFR/IMR) — Invasive physiological measurements are performed using a standard pressure-sensing guidewire.T0 (Acute): FFR, RFR, and IMR are measured in the Non-Culprit Vessel (NCV) and the post-PCI Culprit Vessel (CV).T1 (30-Day): FFR and RFR are measured in the NCV. This T1 pFFR (threshold< 0.80) serves as the gold standard comparator for the primary endpoint.T2 (1-Year): FFR is reassessed in the CV and any untreated NCV.
Diagnostic Test: Cardiac Magnetic Resonance (CMR) — The scan is performed prior to discharge to quantify myocardial injury, including infarct size, Left Ventricular Ejection Fraction (LVEF), and the extent of Microvascular Obstruction (MVO). CMR data serves as the "tissue" component for the secondary 'structure-function-tissue' coupling analysis.

SUMMARY:
Brief Summary The Purpose of the Study : The purpose of this study is to find a safe and reliable "one-stop" solution for treating heart attack patients who have multiple blocked arteries. Currently, doctors face a dilemma: Testing these other blockages during the heart attack procedure is often unreliable.

The most accurate method requires asking the patient to return 30 days later for a second invasive procedure, which is a significant burden.

The Study's Hypothesis : We are testing a new tool called UFR, which uses ultrasound images to measure blockages. Our hypothesis (or "educated guess") is that this new UFR tool is not affected by the body's stress during a heart attack and can provide a true, reliable measurement right away.

The Question the Study is Trying to Answer ： The main question this study is trying to answer is: Can the new "one-stop" UFR tool, used during the initial heart attack procedure, accurately predict which blockages are truly serious... thereby eliminating the need for patients to return for a second procedure 30 days later? Researchers will also follow 200 patients for one year, using advanced scans (like UFR, standard tests, and MRI), to better understand how the heart and arteries heal and change over time.

DETAILED DESCRIPTION:
The ACT-EVOLVE Study: A Prospective, Longitudinal, Multi-modal Study Evaluating the Utility of Acute Phase UFR (IVUS-FFR) to Predict Functional Significance in the Stable Phase for Patients With Acute Coronary Syndrome (ACS).

Study Rationale and Background:

In patients with Acute Coronary Syndrome (ACS) and multi-vessel disease (MVD), complete revascularization (CR) is proven to improve outcomes (e.g., COMPLETE trial, Level A evidence). However, a significant "how-to paradox" exists. Physiologically-guided CR using pressure-wire FFR (pFFR) during the acute index procedure (T0) has failed to show superiority over angiography (e.g., FLOWER-MI trial).This is largely attributed to "functional drift": the acute phase is marked by significant microvascular dysfunction (CMD) and high Index of Microcirculatory Resistance (IMR), especially in STEMI. This interference renders T0 pFFR unreliable, leading to false negatives (over-estimation of FFR).While a staged procedure at a stable timepoint (T1, 30 days) provides a reliable physiological assessment, this strategy faces severe real-world challenges, including high costs, poor patient compliance, and the risk of events during the waiting period.This study hypothesizes that UFR (IVUS-FFR)-a "virtual" FFR derived from IVUS structure and computational fluid dynamics (CFD)-is immune to the acute-phase physiological disturbances (CMD). We hypothesize that T0 UFR can accurately and reliably predict the "gold standard" stable-state pFFR at T1, thus offering a "one-stop shop" solution to guide CR during the index procedure.

Study Objectives:Primary Objective: To assess the diagnostic accuracy (sensitivity, specificity, PPV, NPV, and correlation) of UFR measured in non-culprit vessels (NCV) during the acute phase (T0), compared to the gold-standard pFFR (threshold ≤ 0.80) measured in the stable phase (T1, 30 days).

Key Secondary Objectives:Functional Drift (Head-to-Head): To quantify and compare the "functional re-classification rate" of physiological indices (pFFR, RFR) from T0 to T1 in two pre-specified cohorts: STEMI vs. High-Risk NSTEMI."Structure-Function-Tissue" Coupling (1): To correlate acute culprit vessel (CV) microcirculatory damage (T0 IMR) with sub-acute myocardial tissue injury (MVO and infarct size) measured by T-CMR (3-5 days)."Structure-Function-Tissue" Coupling (2): To analyze the relationship between T0 PCI optimization quality (by post-PCI IVUS criteria) and immediate post-PCI microcirculatory damage (T0 IMR) in the culprit vessel.Longitudinal Vessel Evolution: To assess the long-term (T0 vs. T2) stability of pFFR and UFR in the stented culprit vessel, and to track the functional and structural progression of untreated NCVs (T1 to T2).Prognostic Value: To evaluate the prognostic value of T1 NCV functional status (threshold ≤ 0.80) on 1-year MACE.

Study Design:This is a prospective, longitudinal, observational registry. All key data (physiology, imaging, and CMR) will be analyzed by independent, blinded core laboratories (Physiology Core Lab, Imaging Core Lab, CMR Core Lab). A Clinical Events Committee (CEC) will adjudicate all clinical endpoints.

Study Population:Sample Size: N = 200 patients. Target Population: Patients presenting with ACS (STEMI or High-Risk NSTEMI) who have successfully undergone PCI of the culprit vessel and are found to have MVD.MVD Definition: At least one NCV with a 50-90% diameter stenosis by visual estimation. Pre-specified Stratification:Cohort A: STEMI (N ≈ 100)Cohort B: High-Risk NSTEMI (N ≈ 100)Study Procedures and Timeline:This study involves a systematic, longitudinal assessment at four key timepoints:T0 (Acute Phase - Index Procedure):Culprit Vessel (CV): After successful PCI, post-PCI IVUS, pFFR, RFR, and IMR are measured.Non-Culprit Vessel (NCV): All target NCVs (50-90%) undergo a baseline assessment with IVUS (for UFR calculation) and physiological measurements (T0 pFFR, T0 RFR, T0 IMR).

Key Action: No intervention is performed on the NCV at T0.T-CMR (Sub-Acute Phase - 3-5 Days Post-PCI):Patients (particularly the STEMI cohort) undergo a standardized Cardiac MRI (CMR) to quantify Left Ventricular Ejection Fraction (LVEF), infarct size, and Microvascular Obstruction (MVO).T1 (Stable Phase - 30 Days Post-PCI):Patients return for a planned, invasive follow-up procedure.NCV: The same NCVs assessed at T0 are re-evaluated.Gold Standard Assessment: T1 pFFR and T1 RFR are measured.Clinical Decision: The T1 pFFR result is unblinded. If T1 pFFR threshold ≤ 0.80, the patient undergoes PCI as per guidelines. If > 0.80, the patient continues on optimal medical therapy (OMT).T2 (Long-Term Follow-up - 1 Year):Clinical Follow-up: Assessment for 1-year MACE (cardiac death, target-vessel MI, clinically-driven revascularization).Invasive Follow-up: A planned (per-protocol) 1-year invasive angiographic, IVUS, and functional assessment of both the CV (for in-stent analysis) and any untreated NCV (for disease progression).

Expected Impact:The ACT-EVOLVE registry is designed to provide the first prospective, gold-standard-controlled evidence to validate UFR as a "one-stop" tool for guiding complete revascularization in the acute ACS setting. By directly comparing STEMI and NSTEMI, and building a unique T0-T1-T2 longitudinal database, this study aims to solve the "ultimate dilemma" in ACS-MVD management, potentially replacing the logistically challenging staged-procedure strategy.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years, any sex.
* The participant is able to understand the study procedures and provides voluntary written informed consent.
* Diagnosed with Acute Coronary Syndrome (ACS) and meets the criteria for one of the two pre-specified cohorts:
* STEMI Cohort: Symptom onset < 12 hours with ECG findings of ST-segment elevation myocardial infarction.
* High-Risk NSTEMI Cohort: Meets at least one of the following: GRACE score > 140, dynamic ECG changes (ST-T), or significant Troponin elevation.
* Has undergone successful emergency PCI of the Culprit Vessel (CV), with post-PCI TIMI flow Grade 3.
* Coronary angiography confirms Multi-vessel Disease (MVD), defined as: at least one Non-Culprit Vessel (NCV) with a moderate stenosis (visual diameter stenosis 50-90%).
* The target NCV (50-90% stenosis) is deemed by the investigator to be anatomically suitable for IVUS and pressure-wire assessment.
* The participant agrees and is confirmed to be willing and able to strictly adhere to the protocol and complete all required invasive procedures, CMR scans, and follow-ups at the four timepoints (T0, T-CMR, T1, T2).

Exclusion Criteria:

* Presence of cardiogenic shock on presentation, or persistent hemodynamic instability despite successful PCI of the culprit vessel.
* Known severe allergy to iodinated contrast media or gadolinium-based contrast agents (used for CMR).
* Female participants who are pregnant, breastfeeding, or planning pregnancy within the 1-year study period.Unprotected left main coronary artery disease (stenosis <50%) requiring intervention.
* Prior history of Coronary Artery Bypass Grafting (CABG) surgery.The target NCV has received prior PCI (e.g., existing stent) or surgical revascularization.
* The target NCV is a Chronic Total Occlusion (CTO).
* Severe renal insufficiency (eGFR < 30 ml/min/1.73m²) or currently undergoing chronic dialysis.
* Standard contraindications to CMR examination (e.g., claustrophobia, non-MRI-compatible metallic implants/pacemakers).
* Known presence of a severe non-cardiac comorbidity with an expected lifespan of < 12 months (e.g., advanced malignancy).
* Known severe hematological disease (e.g., severe anemia, active bleeding, thrombocytopenia < 70 x 10⁹/L) rendering the participant unsuitable for multiple invasive procedures.
* Inability to provide informed consent or comply with the complex longitudinal follow-up protocol due to psychiatric, cognitive, or other reasons.
* Currently participating in another interventional (drug or device) clinical study.
* Any other condition which, in the investigator's opinion, makes the participant unsuitable for enrollment (e.g., severe valvular heart disease, cardiomyopathy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be sourced from patients presenting with Acute Coronary Syndrome (STEMI or High-Risk NSTEMI) to the Emergency Department and/or cardiology services of participating multi-center hospitals.
  Eligible participants will be identified and screened for enrollment in the Cardiac Catheterization Laboratory (Cath Lab) immediately following their successful index PCI procedure (T0).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12-02 (Estimated); Primary Completion 2027-06-22 (Estimated); Study Completion 2028-06-22 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Performance of Acute UFR (T0) Compared to Staged pFFR (T1) in Non-Culprit Vessels | Baseline (T0) and 30 Days (T1)
  To assess the diagnostic performance of UFR measured at T0 (Acute) against the gold-standard pFFR (threshold ≤ 0.80) measured at T1 (30 Days). Performance will be assessed by 1) Diagnostic accuracy (Sensitivity, Specificity, PPV, NPV), 2) Correlation (Pearson coefficient and Bland-Altman analysis), and 3) Comparison of Area Under the Curve (AUC).

SECONDARY OUTCOMES:
Functional Re-classification Rate ("Functional Drift") from T0 to T1 (STEMI vs. NSTEMI) | Baseline (T0) and 30 Days (T1)
  To quantify and compare the rate of functional re-classification of pFFR and RFR in the NCV between T0 (Acute) and T1 (Stable). This will be compared head-to-head between the STEMI and High-Risk NSTEMI cohorts.
Correlation between Acute Culprit Vessel IMR and Sub-Acute MVO (Coupling 1) | Baseline (T0) and 3-5 Days (T-CMR)
  To determine the quantitative correlation between the Index of Microcirculatory Resistance (IMR) measured in the Culprit Vessel at T0 and the extent of Microvascular Obstruction (MVO) quantified by Cardiac MRI at T-CMR (3-5 days)
Longitudinal Stability of In-Stent pFFR and UFR (Culprit Vessel Evolution) | Baseline (T0) and 1 Year (T2)
  To compare the temporal stability of pFFR and UFR values measured within the stented segment of the Culprit Vessel from T0 (post-PCI) to T2 (1-year follow-up).
Prognostic Value of T1 NCV Functional Status on 1-Year MACE | From 30 Days (T1) up to 1 Year (T2)
  To evaluate the predictive value of the NCV's functional status at T1 (pFFR ≤ 0.80) on 1-year Major Adverse Cardiovascular Events (MACE). MACE is defined as cardiac death, target vessel MI, and clinically-driven revascularization.

CONTACTS AND LOCATIONS:
Overall Officials: Hai Gao, MD, PHD, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share all de-identified individual participant data (IPD) that underlie the results reported in the main publication(s) for this study. This includes all core clinical, laboratory, and follow-up outcome data, as well as all quantitative data derived from the invasive coronary physiology (pFFR/RFR/IMR), IVUS, and Cardiac MRI (IS/MVO) assessments at all timepoints (T0, T-CMR, T1, T2).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 6 months after the date of the primary manuscript publication, and remaining available for 5 years after the final publication of the main study results.
Access Criteria: Access will be granted to qualified, non-commercial scientific researchers from accredited institutions. Requests must be submitted as a detailed research proposal to the Principal Investigator (PI) and will be reviewed by the Study Steering Committee based on scientific merit and alignment with ethical standards. Approved researchers must sign a formal Data Access Agreement that prohibits attempts at re-identification. Data will be provided via a secure, encrypted platform

REFERENCES:
- [Result] Yu W, Tanigaki T, Ding D, Wu P, Du H, Ling L, Huang B, Li G, Yang W, Zhang S, Yan F, Okubo M, Xu B, Matsuo H, Wijns W, Tu S. Accuracy of Intravascular Ultrasound-Based Fractional Flow Reserve in Identifying Hemodynamic Significance of Coronary Stenosis. Circ Cardiovasc Interv. 2021 Feb;14(2):e009840. doi: 10.1161/CIRCINTERVENTIONS.120.009840. Epub 2021 Feb 5. PMID 33541105
- [Result] Nijveldt R, Maeng M, Beijnink CWH, Piek JJ, Al-Lamee RK, Raposo L, Baptista SB, Escaned J, Davies J, Klem I, Yosofi B, van Geuns RM, Frederiksen CA, Jakobsen L, El Barzouhi A, van der Heijden DJ, Ilhan M, Rasoul S, Brinckman S, Saraber C, Jones DA, Petersen SE, Podlesnikar T, Bunc M, Beijk MAM, Piers LH, van Rees JB, Seligman H, Cole G, Iglesias JF, Degrauwe S, van 't Hof AWJ, Lipsic E, Pundziute-do Prado G, Chattranukulchai P, Rodriguez-Palomares JF, Rigger J, Meuwissen M, Kleijn L, Pereira B, Monti L, van der Schaaf RJ, Sanchis J, Belli G, Tijssen JGP, Thim T, van Royen N; iMODERN Investigators. Immediate or Deferred Nonculprit-Lesion PCI in Myocardial Infarction. N Engl J Med. 2025 Oct 28. doi: 10.1056/NEJMoa2512918. Online ahead of print. PMID 41159879
- [Result] Mehta SR, Wood DA, Storey RF, Mehran R, Bainey KR, Nguyen H, Meeks B, Di Pasquale G, Lopez-Sendon J, Faxon DP, Mauri L, Rao SV, Feldman L, Steg PG, Avezum A, Sheth T, Pinilla-Echeverri N, Moreno R, Campo G, Wrigley B, Kedev S, Sutton A, Oliver R, Rodes-Cabau J, Stankovic G, Welsh R, Lavi S, Cantor WJ, Wang J, Nakamya J, Bangdiwala SI, Cairns JA; COMPLETE Trial Steering Committee and Investigators. Complete Revascularization with Multivessel PCI for Myocardial Infarction. N Engl J Med. 2019 Oct 10;381(15):1411-1421. doi: 10.1056/NEJMoa1907775. Epub 2019 Sep 1. PMID 31475795
- [Result] van der Hoeven NW, Janssens GN, de Waard GA, Everaars H, Broyd CJ, Beijnink CWH, van de Ven PM, Nijveldt R, Cook CM, Petraco R, Ten Cate T, von Birgelen C, Escaned J, Davies JE, van Leeuwen MAH, van Royen N. Temporal Changes in Coronary Hyperemic and Resting Hemodynamic Indices in Nonculprit Vessels of Patients With ST-Segment Elevation Myocardial Infarction. JAMA Cardiol. 2019 Aug 1;4(8):736-744. doi: 10.1001/jamacardio.2019.2138. PMID 31268466
- [Result] Puymirat E, Cayla G, Simon T, Steg PG, Montalescot G, Durand-Zaleski I, le Bras A, Gallet R, Khalife K, Morelle JF, Motreff P, Lemesle G, Dillinger JG, Lhermusier T, Silvain J, Roule V, Labeque JN, Range G, Ducrocq G, Cottin Y, Blanchard D, Charles Nelson A, De Bruyne B, Chatellier G, Danchin N; FLOWER-MI Study Investigators. Multivessel PCI Guided by FFR or Angiography for Myocardial Infarction. N Engl J Med. 2021 Jul 22;385(4):297-308. doi: 10.1056/NEJMoa2104650. Epub 2021 May 16. PMID 33999545